CLINICAL TRIAL: NCT03789136
Title: The Effect of Colon Cancer on Muscle Gene Expression, Body Composition, Muscle Function, and Muscle Metabolism
Acronym: COMUNEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Collaborators: Gelderse Vallei Hospital (Other); Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Other Study IDs: NL58188.081.16
Record Dates: First submitted 2018-12-07; First posted 2018-12-28 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Cachexia; Cancer
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary colon cancer
  Interventions: Other: Not applicable, observational study
- Liver metastases
  Interventions: Other: Not applicable, observational study
- Inguinal hernia (control)
  Interventions: Other: Not applicable, observational study
- Abdominal hysterectomy (control)
  Interventions: Other: Not applicable, observational study

INTERVENTIONS:
Other: Not applicable, observational study — Not applicable, observational study

SUMMARY:
Rationale: Cancer cachexia is a complex metabolic syndrome characterized by clinically relevant loss of muscle mass with or without loss of fat mass. To determine how treatment methods can be most effective, full insight in changes in gene expression, body composition, muscle function and muscle metabolism are of great importance.

Objective: Main aim of the study is to investigate the differences in gene expression, body composition, muscle function and muscle metabolism in colon cancer patients compared to controls.

Study design: Observational study Study population: 40 colon cancer patients undergoing a tumor resection (30 primary tumor and 10 liver metastases) and 15 control patients undergoing an inguinal hernia repair (♂, 10) or an abdominal hysterectomy (♀, 5).

Main study parameters/endpoints: Primary study parameter will be gene expression (transcriptomic and polymerase chain reaction analyses of muscle biopsies). Secondary parameters will be body composition (determined in available CT scans and bio impedance analysis and with DEXA), muscle function parameters (grip and knee flexion/extension strength and measured in a biopsy), metabolic markers (measured in fat and muscle biopsies), biochemical markers (measured in blood/serum) and gene expression of fat biopsies.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The investigators expect no additional risk for the subjects due to the proposed measurements. Biopsies will be taken during the planned operation and therefore is not expected to cause a significant increase in burden for the patient. All other measurements are non-invasive, observational measurements with no risk of any harmful side effects.

ELIGIBILITY:
Inclusion Criteria:

* CC patients:

In order to be eligible to participate in this study, a subject must meet all of the following inclusion criteria:

* Diagnosed with primary colon cancer (30) or liver metastases due to colon cancer(10)
* Eligible for a primary tumor or liver metastases resection procedure

  * Controls:
* Eligible for an inguinal hernia repair (♂, 10) or an abdominal hysterectomy (♀, 5)

Exclusion Criteria:

* CC patients:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Having had chemotherapy or an operational procedure of the abdomen in the past 6 months
* Suffering from malabsorption

  * Controls:
* Having had treatment for previous or current tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — For the control group the investigators include men with inguinal hernia and women eligible for abdominal hysterectomy.
Study Population: 40 colon cancer (CC) patients (♀ and ♂) undergoing primary tumor resection operation (30 patients) or liver metastases surgery (10 patients) and 15 control patients undergoing an inguinal hernia repair (♂, 10) or an abdominal hysterectomy (♀, 5) will be included in the study. Since the investigators do not know the number of patients in the colon cancer group willing to cooperate in the study, the investigators decided to take 5 patients of each control group (50% men and women). Note: during the study the investigators see more men than women joining the study so therefore the investigators raised the number of male controls to 10.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle gene expression | Biopsy during surgery
  Muscle gene expression measured by microarray in a muscle biopsy taken from the rectus abdominis

SECONDARY OUTCOMES:
Body composition | Before surgery
  Measured using single slice staining of CT scan made for diagnostic purposes.
Muscle function | Before surgery
  Measured using hand-grip strength
Muscle protein metabolism | Biopsy during surgery
  Measured in a muscle biopsy taken from the rectus abdominis
Adipose tissue gene expression | Biopsy during surgery
  Adipose tissue gene expression measured using PCR or micro-array in abdominal and subcutaneous fat
Cytokine parameters in the blood | Blood taken prior to surgery
  Blood plasma cytokine levels measured using multiplex or similar technique
Micro-nutrient parameters in the blood | Blood taken prior to surgery
  Micro-nutrient levels in the blood measured using LCMS, ELISA or similar techniques
Cholesterol levels in the blood | Blood taken prior to surgery
  Cholesterol levels in the blood measured by GCMS

CONTACTS AND LOCATIONS:
Overall Officials: Klaske van Norren, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Gelderse Vallei Hospital, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No